CLINICAL TRIAL: NCT02102945
Title: CT Perfusion in the Prognostication of Patients in Coma Following Cardiac Arrest- A Pilot Study
Brief Title: Special Imaging Technique to Aid in the Diagnosis of Patients in Coma After Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP2
Record Dates: First submitted 2014-03-28; First posted 2014-04-03 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2022-10

CONDITIONS: Brain Death
Keywords: Computed tomography; Perfusion imaging; Coma; Heart arrest; Brain death
MeSH Terms: conditions — Brain Death; Coma; Heart Arrest | interventions — Cytidine Triphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Computed tomography perfusion (Other): Participants will undergo CT perfusion of the head after cooling following cardiac arrest.
  Interventions: Procedure: Computed tomography perfusion

INTERVENTIONS:
Procedure: Computed tomography perfusion — Computed tomography perfusion of the head

SUMMARY:
In the present pilot study, the investigators propose to determine if performing CT perfusion scans in post-cardiac arrest patients in coma will help prognosticate the outcome in these patients.

DETAILED DESCRIPTION:
Cardiac arrest is common and is associated with poor survival despite intensive medical care. These patients are subjected to cooling therapy to improve neurological outcomes. After cooling these patients are allowed to spontaneously return to normal body temperature. From here on, the outcome of these patients is mainly dependent on a wait and watch approach as the clinical examination of patients in a coma is very limited. Despite these attempts, 41% of these patients die and only 55 % of them have a favourable neurological outcome.

There have been few clinical scoring systems to provide prognosis in the face of a cardiac arrest but none of them address the more serious group- those in coma. For patients in coma, their medications, particularly those that suppress the central nervous system, cause difficulty in their clinical assessment. Multiple ancillary tests, such as routine CT or MRI of brain, do not give any useful prognostic information. We hypothesize that the neurological outcome of patients in coma is mainly dependent on presence of brainstem function.

To the best of our knowledge, no study has addressed the issue of brainstem function in cardiac arrest patients. This may be due to the fact that there was no imaging tool which could confidently depict the function of the brainstem. In a recently performed study in our institution, using CT perfusion technique, we have demonstrated that patients with diffusely impaired brainstem perfusion have poor prognosis and do not survive. This study is already being considered by the World Health Organization for the modification of criteria for the declaration of brain death. We suggest that a similar imaging technique will potentially be useful in prognosticating patients in coma following cardiac arrest.

In the present pilot study, we propose to determine if performing CT perfusion scans in post-cardiac arrest patients in coma will help prognosticate the outcome in these patients. This may potentially help in early withdrawal of care in patients with significantly impaired brainstem function. If so, this will have a significant impact on patient care and can potentially have huge financial implications for the health care system. Such early decision making may also help in organ harvesting in suitable situations. This will potentially improve the quality of life in many other terminally ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (age range: 18-80 years), in a coma for at least 24 hours following cardiac arrest who are admitted to our cardiac intensive care unit and who have recovered body temperature back to normal after being subjected to the therapeutic hypothermia protocol will be included in the study.
* Also included are those patients whose next of kin have provided consent for the study.

Exclusion Criteria:

* patients who are pregnant,
* those with impaired renal function,
* those who have contraindications to the CT contrast media (such as a known allergy or anaphylactic reactions) and
* those who do not provide consent. Pregnant patients will be excluded to avoid any potential adverse effect of radiation from CT perfusion study on the developing foetus. A developing foetus is more vulnerable to radiation when compared to adult patients.

Patients above 80 years will be excluded to avoid age related comorbidities affecting the patients' survival.

We do not see patients below 18 years of age at our institution thus they will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-06-09 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of brainstem function | 1 year
  Clinical evaluation of brainstem function at the end of hospital stay.

SECONDARY OUTCOMES:
Number of adverse events as a measure of safety and tolerability | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jai JS Shankar, MD, DM, Principal Investigator — Queen Elizabeth II Health Sciences Centre, Halifax Infirmary
Locations (1):
- Queen Elizabeth II Health Sciences Centre-Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No